CLINICAL TRIAL: NCT05908032
Title: A Randomized, Double-blind, Placebo-controlled Phase III Study to Evaluate the Efficacy and Safety of CM310 Under Background Treatment in Patients With Seasonal Allergic Rhinitis Inadequately Controlled With Current Recommended Therapies
Brief Title: Study of CM310 in Subjects With Allergic Rhinitis
Acronym: PHECDA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM310-107206
Record Dates: First submitted 2023-06-02; First posted 2023-06-18 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2023-05

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CM310 group (Experimental): Subcutaneous injection， CM310 4ml for first dose and 2ml for following dose
  Interventions: Biological: CM310
- Placebo (Placebo Comparator): Subcutaneous injection，matching placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: CM310 — IL-4Rα monoclonal antibody
  Arms: CM310 group
Biological: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled phase III clinical study aimed at evaluating the efficacy and safety of CM310 in patients with seasonal allergic rhinitis, and observing the quality of life, PK, PD characteristics, and immunogenicity of subjects.

DETAILED DESCRIPTION:
Allergic rhinitis (AR) is a non infectious chronic inflammatory disease of the nasal mucosa that is mainly mediated by immunoglobulin E (IgE) in atopic individuals exposed to allergens.

All participants will receive standard of care treatment as concomitant medications. CM310 or placebo will be administered as add-on therapy.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand the study and voluntarily sign the ICF;
* Males or females, ≥ 18 and ≤ 65 years old;
* Diagnosed SAR according to the Criteria stated in the Chinese Guidelines for the Diagnosis and Treatment of Allergic Rhinitis (2022, Revised Edition), with or without allergic conjunctivitis, and have SAR history in the same pollen season for at least two years;
* Have immunoglobulin E (IgE)-mediated hypersensitivity to at least one pollen allergen in the current environment, as confirmed by the result of the specific IgE test during the screening/run-in period;
* Adequate pollen exposure during the pollen season: Participants are expected to be in the pollen season for the entire study period and have no travel plans to leave the geographic region more than 48 hours. Definition of a pollen season: the beginning of a pollen season is defined as local pollen count of more than 20/1000 mm2 for three consecutive days, and the end of a pollen season is defined as local pollen count of less than 20/1000 mm2 for three consecutive days.
* Prior to screening, the SAR symptoms of participants remained inadequately controlled (at least one moderate or above SAR symptom) after nasal spray corticosteroids or other SAR medications (antihistamines, leukotriene receptor antagonists, etc.) treatment throughout the same pollen season previously;
* The AM iTNSS ≥ 6 points prior to screening; at the baseline visit, the AM iTNSS ≥ 6 points and the average of the last 6 rTNSS scores ≥ 6 points (i.e., 3 AM and 3 PM assessments over the last three 24-hour periods, including the AM assessment at the baseline visit), with nasal congestion ≥ 2 points and one of the three symptoms of rhinorrhea, nasal itching, and sneezing ≥ 2 points;
* Peripheral blood eosinophils count ≥ 0.3×109/L during the screening/run-in period and baseline visit;
* During the screening/run-in period, participants must complete at least 80% of the assessments in the diary card;
* The participants agree to use highly effective contraception methods from signing of the ICF to 3 months after the last dose of the investigational product.

Exclusion Criteria:

* Use of anti-interleukin 4 receptor alpha subunit (IL-4Rα) monoclonal antibody, thymic stromal lymphopoietin (TSLP) monoclonal antibody, anti-IgE monoclonal antibody, other monoclonal antibodies, or other biologics within 10 weeks or 5 half-lives (whichever is longer) prior to the screening visit;
* Use of any investigational product within 4 weeks prior to the screening visit or planning to participate in other clinical studies during this study;
* Use of systemic immunosuppressants (including but not limited to methotrexate, cyclosporine, mycophenolate mofetil, tacrolimus, penicillamine, sulfasalazine, hydroxychloroquine, azathioprine, cyclophosphamide) for the treatment of inflammatory or autoimmune diseases (e.g., rheumatoid arthritis, inflammatory bowel disease, primary biliary cirrhosis, systemic lupus erythematosus, multiple sclerosis, etc.) within 8 weeks or 5 half-lives (whichever is longer) prior to the screening visit;
* Infections requiring treatment with systemic antibacterial, antiviral, antifungal, antiparasitic, or antiprotozoal medications within 7 days prior to the screening visit;
* Received short-medium-acting systemic corticosteroids (SCS, including oral, intravenous, or intramuscular glucocorticoids), systemic traditional Chinese medicine preparations for the treatment of allergic rhinitis within 4 weeks prior to screening, or long-acting SCS (such as triamcinolone acetonide injection) within 6 weeks prior to screening, or planning to receive the above drugs during the study;
* Use of monoamine oxidase inhibitors within 14 days prior to the screening visit;
* Participants who initiate immunotherapy within 4 weeks prior to the screening visit, or who plan to initiate immunotherapy during the study; Participants who have been receiving immunotherapy at a stable dose within 4 weeks prior to the screening visit and are able to remain this fixed dose throughout the study can be enrolled;
* Participants with concomitant asthma who start treatment with inhaled corticosteroids within 4 weeks prior to screening: Participants who have been treated with a stable dose of inhaled glucocorticoids (≤ 1000 μg/day of fluticasone propionate or equivalent dose of other inhaled glucocorticoids) for at least 4 weeks prior to screening and the dose remains unchanged throughout the study, is in a stable condition at the investigator's discretion, can be enrolled;
* Forced expiratory volume in 1 second (FEV1) ≤ 50% of the predicted value during the screening/run-in period;
* Have active rhinitis of other type except for SAR, such as acute or chronic rhinitis and non-allergic rhinitis;
* Participants with perennial allergic rhinitis (PAR) who are allergic to pet hair. Participants can be enrolled if they stop exposing to pet hair or are allergic to other indoor allergens;
* Patients with active nasal diseases other than SAR, such as acute or chronic rhinosinusitis or nasal septal deviation, which may affect the efficacy evaluation of the investigational product at the investigator's discretion;
* History of any nasal or sinusoidal surgery within 1 year prior to screening;
* Have acute sinusitis, nasal infection, or upper respiratory tract infection at screening or within 2 weeks prior to screening;
* Have benign or malignant tumors in the nasal cavity;
* Previously received an anti-IL-4Rα monoclonal antibody (e.g., dupilumab) for the treatment of AR with poor response (e.g., treatment failure or intolerance);
* Participants who are allergic to MFNS, loratadine, any anti-IL-4Rα monoclonal antibody or any component of CM310;
* Comorbidity of other poorly controlled serious diseases or chronic diseases, including but not limited to active infection, cardiovascular and cerebrovascular diseases, pulmonary tuberculosis or other pathogen infections, diabetes, autoimmune diseases, human immunodeficiency virus infection, treponema pallidum infection, active hepatitis B, hepatitis C or parasitic diseases;
* Participants with malignancy within 5 years prior to screening (except for completely cured cervical carcinoma in situ and non-metastatic squamous cell or basal cell carcinoma of the skin);
* Participants with severe hepatic or renal impairment, such as aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2 times the upper limit of normal (ULN), total bilirubin > 1.5 times the ULN, or serum creatinine > 1.2 times the ULN;
* Have received a live-attenuated vaccine within 12 weeks prior to randomization or planning to receive one during the study;
* Known or suspected immunosuppression, including but not limited to a history of invasive opportunistic infections (eg, tuberculosis, histoplasmosis, listeriosis, coccidioidomycosis, pneumocystosis, aspergillosis), even after this infection condition has recovered; or with unusually frequent, recurrent, or long-term infections at the investigator's discretion;
* Pregnant or breast-feeding women, or women who plan to become pregnant or breast-feeding during the study;
* Heavy alcohol consumption [i.e., more than 14 units of alcohol per week (1 unit = 360 mL of beer or 45 mL of distilled spirits with 40% alcohol or 150 mL of wine)] or history of drug abuse within 3 months prior to screening;
* Participants with any other conditions that are considered by the investigator as unsuitable to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2023-12-04 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in daily reflective total nasal symptom scores (rTNSS) over 2 weeks of treatment. | Up to week 4
  The total nasal symptom score (TNSS) is the sum of the four symptom scores for rhinorrhea, nasal congestion, nasal itching, and sneezing, where each symptom is scored on a scale of 0 to 3.

SECONDARY OUTCOMES:
Mean change from baseline in daily rTNSS over 4 weeks of treatment | Up to week 4
  The total nasal symptom score (TNSS) is the sum of the four symptom scores for rhinorrhea, nasal congestion, nasal itching, and sneezing, where each symptom is scored on a scale of 0 to 3.
Mean change from baseline in the daily AM and PM reflective total nasal symptom score (AM and PM rTNSS) over 2 and 4 weeks of treatment | Up to week 4
  The total nasal symptom score (TNSS) is the sum of the four symptom scores for rhinorrhea, nasal congestion, nasal itching, and sneezing, where each symptom is scored on a scale of 0 to 3.
Mean change and mean percent change from baseline in daily AM pre-dose instantaneous total nasal symptom score (iTNSS) over 2 weeks and 4 weeks of treatment | Up to week 4
  The instantaneous total symptom scores (iTNSS) are the rating of the severity of instantaneous symptoms at a time point.
Mean percent change from baseline in daily rTNSS over 2 and 4 weeks of treatment | Up to week 4
  The total nasal symptom score (TNSS) is the sum of the four symptom scores for rhinorrhea, nasal congestion, nasal itching, and sneezing, where each symptom is scored on a scale of 0 to 3.
Mean change from baseline in daily rTNSS (including AM rTNSS and PM rTNSS) for individual nasal symptoms (rhinorrhea, nasal congestion, nasal itching, and sneezing) over 2 and 4 weeks of treatment | Up to week 4
  The total nasal symptom score (TNSS) is the sum of the four symptom scores for rhinorrhea, nasal congestion, nasal itching, and sneezing, where each symptom is scored on a scale of 0 to 3.
Mean change and mean percent change from baseline in daily reflective total ocular symptom score (rTOSS) over 2 weeks or 4 weeks of treatment | Up to week 4
  The total ocular symptom score (TOSS) is the sum of three symptom scores for itchy/burning eyes, watery eyes, and red eyes, where each symptom is scored on a scale of 0 to 3.
Mean change from baseline in daily AM and PM reflective total ocular symptom score (AM and PM rTOSS) over 2 weeks and 4 weeks of treatment | Up to week 4
  The total ocular symptom score (TOSS) is the sum of three symptom scores for itchy/burning eyes, watery eyes, and red eyes, where each symptom is scored on a scale of 0 to 3.
Mean change from baseline in daily AM pre-dose instantaneous total ocular symptom score (iTOSS) over 2 weeks and 4 weeks of treatment | Up to week 4
  The instantaneous total symptom scores (iTOSS) are the rating of the severity of instantaneous symptoms at a time point.
Mean percent change from baseline in daily rTOSS over 2 weeks and 4 weeks of treatment | Up to week 4
  The total ocular symptom score (TOSS) is the sum of three symptom scores for itchy/burning eyes, watery eyes, and red eyes, where each symptom is scored on a scale of 0 to 3.
Mean percent change from baseline in daily AM pre-dose iTOSS over 2 weeks and 4 weeks of treatment | Up to week 4
  The instantaneous total symptom scores (iTOSS) are the rating of the severity of instantaneous symptoms at a time point.
Mean change from baseline in daily rTOSS (including AM and PM rTOSS) for individual symptoms (itching/burning eyes, tearing/watering eyes, and eye redness) over 2 weeks and 4 weeks of treatment | Up to week 4
  The total ocular symptom score (TOSS) is the sum of three symptom scores for itchy/burning eyes, watery eyes, and red eyes, where each symptom is scored on a scale of 0 to 3.
The change from baseline in rhinoconjunctivitis quality of life questionnaire (RQLQ) score in allergic rhinitis participants over 2 weeks and 4 weeks of treatment | Up to week 4
  The Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) is a 28-item, self-administered, disease-specific (AR) quality of life scale used by participants to assess quality of life over a week.
Time to onset of treatment effect | Up to week 4
  The reflective scores (rTNSS, rTOSS) represent the participant's symptoms in the previous 12 hours. The instantaneous total symptom scores (iTNSS, iTOSS) are the rating of the severity of instantaneous symptoms at a time point.
Time to maximum treatment effect | Up to week 4
  The reflective scores (rTNSS, rTOSS) represent the participant's symptoms in the previous 12 hours. The instantaneous total symptom scores (iTNSS, iTOSS) are the rating of the severity of instantaneous symptoms at a time point.
Area under the curve of the change from baseline in the daily rTNSS over 2 weeks and 4 weeks of treatment | Up to week 4
  The total nasal symptom score (TNSS) is the sum of the four symptom scores for rhinorrhea, nasal congestion, nasal itching, and sneezing, where each symptom is scored on a scale of 0 to 3.
Number of days with no or mild symptoms over 2 weeks and 4 weeks of treatment | Up to week 4
  Based on all the endpoints of TNSS and TOSS.
Incidence of adverse events (AEs) | Up to wee 12
  Evaluate the incidence of treatment-emergency adverse events.
Serum CM310 concentration | Up to week 12
  Collect the blood samples for Pharmacokinetics analysis
Change and percent change from baseline of human thymus and activation-regulated chemokine (TARC) | Up to week 12
  Collect the blood samples for Pharmacodynamics analysis
change and percent change from baseline of total immunoglobulin E (IgE) in serum/plasma | Up to week 12
  Collect the blood samples for Pharmacodynamics analysis
change and percent change from baseline of counts and ratios of eosinophil in blood | Up to week 12
  Collect the blood samples for Pharmacodynamics analysis
The development of anti-drug antibody (ADA) and neutralizing antibody (Nab) | Up to week 12
  Collect the blood samples for anti-drug antibody testing

CONTACTS AND LOCATIONS:
Overall Officials: Luo Zhang, Principal Investigator — Beijing Tong-Ren hospital
Locations (1):
- Beijing Tong-Ren hospital, Beijing, China

REFERENCES:
- [Derived] Zhang Y, Li J, Wang M, Li X, Yan B, Liu J, Shi L, Cao Z, Feng Y, Liu W, Xu Z, Ma R, Gao X, Liu W, Xue J, Ren X, Li X, Song X, Yang Y, Wang Y, Xing Z, Quan F, Pan J, Sun Y, Shi F, Chen X, Yan H, Zhao G, Chen B, Wang C, Zhang L. Stapokibart for moderate-to-severe seasonal allergic rhinitis: a randomized phase 3 trial. Nat Med. 2025 Jul;31(7):2213-2221. doi: 10.1038/s41591-025-03651-5. Epub 2025 Apr 4. PMID 40186079
- [Derived] Wang M, Zhang Y, Li J, Wang C, Zhang L. Stapokibart (CM310) in patients with uncontrolled seasonal allergic rhinitis (PHECDA): Rationale and design of a multicentre, randomized, double-blind, placebo-controlled study. Asia Pac Allergy. 2025 Mar;15(1):15-20. doi: 10.5415/apallergy.0000000000000174. Epub 2025 Jan 13. PMID 40051426
- [Derived] Zhang Y, Yan B, Zhu Z, Wang X, Song X, Zhu D, Ma T, Zhang Y, Meng C, Wang G, Wang C, Zhang L. Efficacy and safety of stapokibart (CM310) in uncontrolled seasonal allergic rhinitis (MERAK): an investigator-initiated, placebo-controlled, randomised, double-blind, phase 2 trial. EClinicalMedicine. 2024 Feb 6;69:102467. doi: 10.1016/j.eclinm.2024.102467. eCollection 2024 Mar. PMID 38356731